CLINICAL TRIAL: NCT02972437
Title: Detection of Group A Streptococcus (GAS) in Oral Cavity Using Molecular Techniques
Brief Title: Detection of Group A Streptococcus (GAS) in Oral Cavity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: naamap-HMO-CTIL
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Tonsillitis
Keywords: GAS in oral cavity
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: sample taking — throat culture and oral cavity sample

SUMMARY:
The investigators intend to screen children who are suspected of having GAS tonsillitis. From each child we will take a throat culture and saliva sample to screen for molecular evidence of GAS.

ELIGIBILITY:
Inclusion Criteria:

* clinical evidence of GAS tonsillitis
* healthy, no chronic illness
* not a GAS carrier

Exclusion Criteria:

* GAS carrier
* Active background disease

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children 3-16 years old with evidence of tonsilitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
molecular detection of GAS compared to throat culture detection | 3 days
  3 days after taking the oral sample, the investigators will compare it to the throat culture taken at the same time.

IPD SHARING:
Plan to Share IPD: No